CLINICAL TRIAL: NCT07299435
Title: Effect of the Combination of Dexamethasone and BIS Monitoring on Reducing Postoperative Nausea and Vomiting in Children: a Multicenter Prospective Double-blind Study (BISDEX TRIAL)
Brief Title: Effect of the Combination of Dexamethasone and BIS Monitoring on Reducing Postoperative Nausea and Vomiting in Children
Acronym: BISDEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: Municipal Hospital Ostrava (Other); Havířov Hospital (Unknown); Frýdek-Místek Hospital (Unknown); Tomas Bata Hospital, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FNO-KARIM-BISDEX
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Tonsil Hypertrophy
Keywords: postoperative nausea and vomiting; emergence delirium; children; ENT surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group - BIS monitoring (Experimental): Following the administration of dexamethasone, BIS monitoring will be initiated immediately, with the depth of general anaesthesia controlled to a BIS value of 40-60.
  Interventions: Procedure: BIS monitoring
- Control group - sham BIS monitoring (Experimental): A non-functional electrode for bispectral index (BIS) monitoring will then be attached to the patient's forehead. The depth of anaesthesia will be controlled based on the minimum alveolar concentration (target MAC: 1-1.1).
  Interventions: Procedure: Sham BIS monitoring

INTERVENTIONS:
Procedure: BIS monitoring — BIS monitoring will be used to guide the depth of anaesthesia in this intervention group.
  Arms: Intervention group - BIS monitoring
Procedure: Sham BIS monitoring — Sham BIS monitoring will be used in this control group, the depth of anaesthesia will be guided by the values of minimum alveolar concentration.
  Arms: Control group - sham BIS monitoring

SUMMARY:
This study will investigate the impact of combining dexamethasone and bispectral index (BIS) monitoring on the incidence of postoperative nausea and vomiting, emergence delirium and recovery trajectories in children undergoing ear-nose-throat (ENT) surgery.

DETAILED DESCRIPTION:
Immediately after securing the airway, an electrode will be attached and BIS monitoring will begin. This will be used to control the depth of general anaesthesia throughout the entire surgical procedure, with the aim of achieving BIS values of 40-60.

Intervention group: Following the administration of dexamethasone at the same dos-age as in the control group, BIS monitoring will be initiated immediately, with the depth of general anaesthesia controlled to a BIS value of 40-60.

Control group: Once access to the vascular system has been secured, dexamethasone will be administered intravenously at a dose of 0.15 mg/kg body weight, up to a maxi-mum of 5 mg. A non-functional electrode for bispectral index (BIS) monitoring will then be attached to the patient's forehead. The depth of anaesthesia will be controlled based on the minimum alveolar concentration (target MAC: 1-1.1).

ELIGIBILITY:
Inclusion Criteria:

* children aged 2 to 8 years undergoing endoscopic adenoidectomy
* parental/child consent
* ASA I-II (American Society of Anaesthesiologists Physical Status)
* no central nervous system (CNS) or gastrointestinal tract (GIT) disease
* no corticosteroid medication

Exclusion Criteria:

* Parent/child disapproval
* ASA III and above (American Society of Anaesthesiologists Physical Status)
* central nervous system (CNS) or gastrointestinal tract (GIT) disease
* chronic corticosteroid therapy

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1508 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Effect of BIS monitoring on the incidence of postoperative nausea and vomiting | 24 hours
  Effect of BIS monitoring on the incidence of postoperative nausea and vomiting within 24 hours after surgery under general anaesthesia. Vomiting is defined as the expulsion of gastric contents through the oral cavity. Nausea is defined for the purposes of this study using the Baxter Animated Retching Face (BARF) score of 4 or more.

SECONDARY OUTCOMES:
Effect of BIS monitoring on the incidence of emergent delirium | 1 hour from surgery
  Effect of BIS monitoring on the incidence of emergent delirium (Paediatric Anaesthesia Emergence Delirium (PAED) above 10 and Watcha scale above 3) in the PACU.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Frelich, MD, Ph.D., Principal Investigator — University Hospital Ostrava
Locations (5):
- Czechia (5):
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - Frýdek-Místek Hospital, Frýdek-Místek
  - Havířov Hospital, Havířov
  - Municipal Hospital Ostrava, Ostrava
  - Tomáš Baťa Hospital, Zlín, Zlín

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon reasonable request.